CLINICAL TRIAL: NCT00761150
Title: A Phase 3, Open-Label Period Followed by a Randomized, Double-blind, Placebo-controlled Study of the Analgesic Efficacy of Extended-release Hydrocodone/Acetaminophen (Vicodin CR) Compared to Placebo in Subjects With Chronic Low Back Pain
Brief Title: Study to Evaluate the Safety and Efficacy of ABT-712 in Subjects With Moderate to Severe Chronic Low Back Pain (CLBP)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: AbbVie (prior sponsor, Abbott) (Industry)
Responsible Party: Sponsor
Organization: AbbVie (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: M10-385
Record Dates: First submitted 2008-09-25; First posted 2008-09-29 (Estimated); Results first posted 2013-12-23 (Estimated); Last update posted 2014-02-07 (Estimated); Status verified 2014-01

CONDITIONS: Chronic Low Back Pain
Keywords: Effect on sleep interference by pain
MeSH Terms: interventions — Hydrocodone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Open-label ABT-712 (Experimental): 2 ABT-712 extended-release tablets, twice daily, for up to 3 weeks (open-label period).
  Interventions: Drug: ABT-712
- Double-blind ABT-712 (Experimental): 2 ABT-712 extended-release tablets, twice daily, for 4 weeks (double-blind period).
  Interventions: Drug: ABT-712
- Double-blind Placebo (Placebo Comparator): 2 placebo tablets, twice daily, for 4 weeks (double-blind period).
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: ABT-712 — ABT-712 extended-release tablet
  Other Names: Hydrocodone and acetaminophen extended-release; Hydrocodone bitartrate and acetaminophen extended-release
  Arms: Double-blind ABT-712; Open-label ABT-712
Drug: Placebo — Placebo tablet
  Arms: Double-blind Placebo

SUMMARY:
The primary purpose of the study was to test the efficacy of 2 tablets (twice daily) of ABT-712, compared to placebo, administered over a 4-week period in participants with moderate to severe mechanical chronic low back pain (CLBP).

DETAILED DESCRIPTION:
The study used a randomized withdrawal design with an open label (OL) period prior to a double-blind (DB) period. Participants who were receiving benefit and were tolerating ABT-712 during the OL period were randomized into the DB period. Study drug was given for a total of 8 weeks, which included up to 3 weeks in OL, up to 4 weeks in DB, and a 1-week DB taper. During the OL period, all participants took increasing doses of ABT-712 until they were taking 2 tablets, twice daily. During the DB period, participants in the ABT-712 group took 2 ABT-712 tablets, twice daily throughout the 4 weeks, while participants in the placebo group took 2 placebo tablets twice daily.

ELIGIBILITY:
Inclusion Criteria:

* Adult male and female subjects who voluntarily sign the informed consent
* Diagnosis of CLBP of 6 months duration

Exclusion Criteria:

* Incapacitated or bedridden subjects
* Subjects with history of surgical or invasive intervention

Ages: 21 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 308 (Actual)
Dates: Start 2008-09; Primary Completion 2009-03 (Actual); Study Completion 2009-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pedro Quintana Diez, MD, Study Director — AbbVie
Locations (32):
- United States (32):
  - Site Reference ID/Investigator# 10143, Tempe, Arizona
  - Site Reference ID/Investigator# 10161, Tempe, Arizona
  - Site Reference ID/Investigator# 10155, Tucson, Arizona
  - Site Reference ID/Investigator# 10160, Anaheim, California
  - Site Reference ID/Investigator# 10821, Lomita, California
  - Site Reference ID/Investigator# 10152, Clearwater, Florida
  - Site Reference ID/Investigator# 10157, DeLand, Florida
  - Site Reference ID/Investigator# 10142, Oldsmar, Florida
  - Site Reference ID/Investigator# 10147, Pembroke Pines, Florida
  - Site Reference ID/Investigator# 13821, Plantation, Florida
  - Site Reference ID/Investigator# 15821, Chicago, Illinois
  - Site Reference ID/Investigator# 10136, Crestview Hills, Kentucky
  - Site Reference ID/Investigator# 10822, New Orleans, Louisiana
  - Site Reference ID/Investigator# 10140, Shreveport, Louisiana
  - Site Reference ID/Investigator# 10158, Brockton, Massachusetts
  - Site Reference ID/Investigator# 13601, Fall River, Massachusetts
  - Site Reference ID/Investigator# 10162, Wellesley Hills, Massachusetts
  - Site Reference ID/Investigator# 10159, Omaha, Nebraska
  - Site Reference ID/Investigator# 10126, Las Vegas, Nevada
  - Site Reference ID/Investigator# 10156, Cincinnati, Ohio
  - Site Reference ID/Investigator# 10148, Cincinnati, Ohio
  - Site Reference ID/Investigator# 10151, Kettering, Ohio
  - Site Reference ID/Investigator# 10138, Marion, Ohio
  - Site Reference ID/Investigator# 10150, Perrysburg, Ohio
  - Site Reference ID/Investigator# 10141, Dallas, Texas
  - Site Reference ID/Investigator# 10149, El Paso, Texas
  - Site Reference ID/Investigator# 10130, Fort Worth, Texas
  - Site Reference ID/Investigator# 10163, Killeen, Texas
  - Site Reference ID/Investigator# 13201, San Antonio, Texas
  - Site Reference ID/Investigator# 10154, San Antonio, Texas
  - Site Reference ID/Investigator# 10144, Roanoke, Virginia
  - Site Reference ID/Investigator# 10113, Spokane, Washington

REFERENCES:
- See also: Related Info — http://rxabbvie.com

RESULTS

PARTICIPANT FLOW:
Period: Open-label Period
Arm/Group | Open-label ABT-712 | Double-blind ABT-712 | Double-blind Placebo
Started | 308 | 0 | 0
Completed | 238 | 0 | 0
Not Completed | 70 | 0 | 0
Not completed — Adverse Event | 36 | 0 | 0
Not completed — Did not meet DB randomization criteria | 11 | 0 | 0
Not completed — Lost to Follow-up | 7 | 0 | 0
Not completed — Lack of Efficacy | 4 | 0 | 0
Not completed — Withdrawal by Subject | 5 | 0 | 0
Not completed — Noncompliance | 2 | 0 | 0
Not completed — Other | 5 | 0 | 0
Period: Double-blind Period
Arm/Group | Open-label ABT-712 | Double-blind ABT-712 | Double-blind Placebo
Started | 0 | 120 | 118
Completed | 0 | 106 | 89
Not Completed | 0 | 14 | 29
Not completed — Lack of Efficacy | 0 | 2 | 19
Not completed — Adverse Event | 0 | 3 | 3
Not completed — Withdrawal by Subject | 0 | 3 | 2
Not completed — Lost to Follow-up | 0 | 2 | 1
Not completed — Did not meet DB randomization criteria | 0 | 0 | 1
Not completed — Noncompliance | 0 | 1 | 0
Not completed — Other | 0 | 3 | 3

BASELINE CHARACTERISTICS:
Groups:
- Nonrandomized: 2 ABT-712 extended-release tablets, twice daily, for up to 3 weeks during the open-label period. These participants enrolled in the study and received at least 1 dose of study drug, and either discontinued during the open-label period or were not randomized and did not progress to the double-blind period.
- Total: Total of all reporting groups
Arm/Group | Nonrandomized | Double-blind ABT-712 | Double-blind Placebo | Total
Number analyzed (Participants) | 70 | 120 | 118 | 308
Age, Continuous [Mean (Standard Deviation); unit: years] | 51.3 (12.31) | 48.1 (12.64) | 48.4 (12.24) | 49.0 (12.44)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 43 | 66 | 78 | 187
  Male | 27 | 54 | 40 | 121
Double-blind Baseline CLBP Intensity VAS [Mean (Standard Deviation); unit: scores on a scale] — The last assessment using the CLBP Intensity Visual Analog Scale (VAS) (0 mm = No Pain and 100 mm = Worst Pain Imaginable) conducted before the first dose in the double-blind period.
  scores on a scale | NA (NA) — These subjects were not randomized to the double-blind period. | 22.4 (15.25) | 22.9 (14.86) | 22.6 (15.03)
Double-blind Baseline Sleep Interference by Pain Scale [Mean (Standard Deviation); unit: scores on a scale] — The last assessment of how much back pain interfered with their sleep on a scale of 0 (not at all) to 10 (completely) conducted before the first dose in the double-blind period.
  scores on a scale | NA (NA) — These subjects were not randomized to the double-blind period. | 2.2 (2.01) | 2.1 (1.82) | 2.2 (1.91)

OUTCOME MEASURES:

1. Primary Outcome: Change From Double-blind (DB) Baseline to Final Assessment in Chronic Lower Back Pain (CLBP) Intensity by Visual Analog Scale (VAS)
Description: The change from the DB randomization baseline (DB baseline: the last assessment before first dose in the DB period) to the final assessment in pain intensity, assessed using the CLBP Intensity VAS (0 mm = No Pain and 100 mm = Worst Pain Imaginable). Least squares means and standard errors from 2-way ANCOVA model without interaction.
Time Frame: Double-blind baseline to 4 weeks
Population: The analysis of the primary outcome measure included all randomized participants who received at least 1 dose of study drug during the double-blind period (double-blind intent-to-treat).
Measure: Least Squares Mean (Standard Error); unit: scores on a scale
Arm/Group | Double-blind ABT-712 | Double-blind Placebo
Number analyzed (Participants) | 120 | 118
scores on a scale | 1.1 (2.41) | 18.0 (2.43)

2. Secondary Outcome: Change From Double-blind (DB) Baseline to Final Assessment in Chronic Pain Sleep Inventory (CPSI)
Description: The change from the DB randomization baseline (DB baseline: the last assessment before first dose in the DB period) to the final assessment of the impact of pain on the participant's sleep. The CPSI utilizes a 100 mm VAS scale for questions of how often the participant had trouble falling asleep because of pain, needed sleeping medication, was awakened by pain during the night, and was awakened by pain in the morning (0 mm = Never and 100 mm = Always); and for rating the overall quality of sleep (0 mm = Very Poor and 100 mm = Excellent). Least squares means and standard errors from 2-way ANCOVA model without interaction.
Time Frame: Double-blind baseline to 4 weeks
Population: The analysis of the secondary outcome measure included all randomized participants who received at least 1 dose of study drug during the DB period (DB intent-to-treat), had a DB baseline assessment, and had at least 1 assessment during the DB period.
Measure: Least Squares Mean (Standard Error); unit: scores on a scale
Arm/Group | Double-blind ABT-712 | Double-blind Placebo
Number analyzed (Participants) | 116 | 113
scores on a scale
  Trouble Falling Asleep | -4.8 (2.43) | 13.1 (2.48)
  Needed Sleeping Medication | -1.6 (2.04) | 8.4 (2.09)
  Awakened by Pain During the Night | -0.5 (2.52) | 15.1 (2.57)
  Awakened by Pain in the Morning | 0.3 (2.62) | 13.0 (2.67)
  Quality of Sleep | 0.1 (2.59) | -13.9 (2.66)

ADVERSE EVENTS:
Time Frame: AEs were recorded from the time of study drug administration to 30 days after last dose (total 12 weeks); SAEs were recorded from the time that informed consent was obtained until 30 days following discontinuation of study drug (total 16 weeks).
Description: AEs with onset during the OL period are shown separately from AEs with onset after the first dose of study drug (ABT-712 or placebo) in the DB period.
Arm/Group | Open-label ABT-712 | Double-blind ABT-712 | Double-blind Placebo
Serious Adverse Events (participants affected / at risk) | 1/308 | 0/120 | 2/118
Other Adverse Events (participants affected / at risk) | 169/308 | 18/120 | 19/118
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Open-label ABT-712 (N=308) | Double-blind ABT-712 (N=120) | Double-blind Placebo (N=118)
DIVERTICULAR PERFORATION (Gastrointestinal disorders) | 1 | 0 | 0
ANXIETY (Psychiatric disorders) | 0 | 0 | 1
DEPRESSION (Psychiatric disorders) | 0 | 0 | 1
PULMONARY EMBOLISM (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Open-label ABT-712 (N=308) | Double-blind ABT-712 (N=120) | Double-blind Placebo (N=118)
CONSTIPATION (Gastrointestinal disorders) | 84 | 5 | 4
NAUSEA (Gastrointestinal disorders) | 78 | 8 | 2
VOMITING (Gastrointestinal disorders) | 21 | 4 | 2
DIZZINESS (Nervous system disorders) | 23 | 1 | 2
HEADACHE (Nervous system disorders) | 28 | 7 | 13
SOMNOLENCE (Nervous system disorders) | 32 | 1 | 1
PRURITUS (Skin and subcutaneous tissue disorders) | 20 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
AbbVie requests that any investigator or institution that plans on presenting/publishing results disclosure, provide written notification of their request 60 days prior to their presentation/publication. AbbVie requests that no presentation/publication will be instituted until 12 months after a study is completed, or after the first presentation/publication whichever occurs first. A delay may be proposed of a presentation/publication if AbbVie needs to secure patent or proprietary protection.